CLINICAL TRIAL: NCT05964322
Title: Cardiac Rehabilitation of Children and Adolescent With Long QT Syndrome
Acronym: RYTHMO'FIT
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: RECHMPL23_0225
Record Dates: First submitted 2023-07-04; First posted 2023-07-27 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Long QT Syndrome; Congenital Long Qt Syndrome; Inherited Cardiac Conduction Disorder; Pediatric ALL
Keywords: Cardiac Rehabilitation; Long QT syndrome; Pediatric; Exercise training; Educational program
MeSH Terms: conditions — Long QT Syndrome; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Children and adolescents with inherited cardiac arrhythmia su ch Long QT Syndrome (LQTS) have lower physical and quality of life than their healthy peers. A multi-component cardiac rehabilitation, including an exercise training program and education program, might counteract those effects.

The goal of this pilot study is to evaluate the security, feasibility, and benefits of a cardiac rehabilitation program in children with LQTS aged between 6 to 18 years old.

The main question[s] it aims to answer are:

* Is center-based cardiac rehabilitation safe and feasible for children with LQTS?
* Does a 12-week cardiac rehabilitation program improve physical fitness and quality of life?

DETAILED DESCRIPTION:
Physical fitness is an independent predictor of all-cause mortality and global health in the general population. Assessments of cardiorespiratory and muscle fitness in children with chronic illness are growing in interest, even in less prevalent chronic diseases. For instance, children and adolescents with Long QT Syndrome (LQTS) have lower cardiorespiratory fitness, muscle strength, and quality of life than their healthy peers.

A multi-component cardiac rehabilitation including an exercise training program and education program might counteract this lowered physical fitness.

The RYTHMO'FIT pilot study seeks to test the security, and feasibility, and to evaluate the benefits of an innovative center-based program to improve physical and mental health in children and adolescents with LQTS.

In this retrospective study, eight children had undergone a 12-week program, within each session composed by:

* A 1-hour exercise training session with a trained exercise physiologist: resistance training, aerobic training, stretching, and different activity (e.g., basketball, handball, football, hockey)
* A 30-min educational workshop with a specialist nurse (e.g., beta-blockade, sports participation, healthy behaviors).
* A 10-min medical interview with a cardiologist to have feedback from parents and patients on each session and the past 7 seven days.

We hypothesized the RYTHMO'FIT study is safe, feasible, and provides benefits for mental and physical health in children and adolescents with LQTS. If the results of this pilot study are positive, they will lead to a larger randomized multicentric controlled trial to evaluate the effectiveness of a hybrid cardiac rehabilitation program in children, adolescents, and young adults with LQTS.

ELIGIBILITY:
* Children and adolescents, aged 6 to 18 years old, diagnosed with congenital LQTS and had been recently under medical check-up in our last study QUALIMYORYTHM
* With impaired cardiorespiratory fitness (VO2 peak <80% of predicted values or VAT <55% of predicted values) or with normal cardiorespiratory fitness but requiring patient education and information on limits/security in taking part in sports participation.
* Willingness and ability for parents and children to take part in a 12-week center-based program (e.g., availability during the school period, transportation options)
* Informed consent of parents or legal guardians, and oral assent of children.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children aged 8 to 18 years with an LQTS.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Security | At week 12
  Count and specify any cardiac events on the ECG scope during each session. Reporting of related and non-related event during the past 7 days through short questionnaire each week.
Recruitment rates | At week 12
  Number of participants who completed baseline assessment compared to the number who were eligible (expressed in %).
Retention rates | At week 12
  Participants who participated in the 12-week intervention and completed the follow-up assessments at the end of the program (expressed in %).
Adherence | At week 12
  Percentage exercise sessions attained by participants compared to number of sessions proposed.

SECONDARY OUTCOMES:
Change on cardiorespiratory fitness | between week 0 and week 12
  Assessing the following variables by cardiopulmonary exercise testing: peak oxygen uptake (VO2peak), ventilatory anaerobic threshold (VAT), ventilatory efficiency (VE/VCO2 slope), maximum heart rate (HR), oxygen pulse (VO2/HR), maximal power, respiratory exchange ratio.
Change on muscle architecture | between week 0 and week 12
  Assessing the following variables by ultrasounding: Anatomical cross sectional area, pennation angle, fascicle length and muscle thickness
Change on muscle strength | between week 0 and week 12
  Lower and upper limb maximal isometric strength by knee extension and handgrip test, respectively. Lower body explosive muscular strength was assessed by standing long broad jump.
Change on physical activity level | between week 0 and week 12
  Time spent in vigorous, moderate-to-vigorous, light physical activity assessed by waist-worn tri axial accelerometer during 7 days.
Change on Self reported total score of the Pediatric Quality of Life Inventory (PedsQL) 4.0 questionnaire | between week 0 and week 12
Change on Proxy-reported total score of the Pediatric Quality of Life Inventory (PedsQL) | between week 0 and week 12
Pediatric Quality of Life Inventory (PedsQL) 4.0 Health-related quality (HRQoL ) of life questionnaire score per dimension (self and proxy reports) | between week 0 and week 12
Change on cardiological outcomes | between week 0 and week 12
  Electrocardiographic at rest (QTc, heart rate, PR, QRS interval time) and echocardiography (LVEF, IVSd, IVSs, LVEDV, E/A ratio)

CONTACTS AND LOCATIONS:
Overall Officials: Pascal AMEDRO, Professor, Principal Investigator — University Hospital of Bordeaux - Haut-Levêque Hospital
Locations (2):
- France (2):
  - University Hospital of Montpellier - Arnaud de Villeneuve Hospita, Montpellier
  - Saint-Pierre Institute, Palavas-les-Flots

REFERENCES:
- [Background] Souilla L, Avesani M, Boisson A, Requirand A, Matecki S, Vincenti M, Werner O, De La Villeon G, Pommier V, Pasquie JL, Guillaumont S, Amedro P. Cardiorespiratory fitness, muscle fitness, and physical activity in children with long QT syndrome: A prospective controlled study. Front Cardiovasc Med. 2023 Jan 11;9:1081106. doi: 10.3389/fcvm.2022.1081106. eCollection 2022. PMID 36712265
- [Background] Amedro P, Werner O, Abassi H, Boisson A, Souilla L, Guillaumont S, Calderon J, Requirand A, Vincenti M, Pommier V, Matecki S, De La Villeon G, Lavastre K, Lacampagne A, Picot MC, Beyler C, Delclaux C, Dulac Y, Guitarte A, Charron P, Denjoy-Urbain I, Probst V, Baruteau AE, Chevalier P, Di Filippo S, Thambo JB, Bonnet D, Pasquie JL. Health-related quality of life and physical activity in children with inherited cardiac arrhythmia or inherited cardiomyopathy: the prospective multicentre controlled QUALIMYORYTHM study rationale, design and methods. Health Qual Life Outcomes. 2021 Jul 28;19(1):187. doi: 10.1186/s12955-021-01825-6. PMID 34321045
- [Result] Souilla L, Guillaumont S, Auer A, Metzler G, Requirand A, Vincenti M, De La Villeon G, Pasquie JL, Mottet D, Amedro P. Cardiac rehabilitation in children and adolescents with long QT syndrome: the RYTHMO'FIT pilot study. BMC Sports Sci Med Rehabil. 2024 Jul 12;16(1):152. doi: 10.1186/s13102-024-00941-2. PMID 38997778